CLINICAL TRIAL: NCT05226325
Title: Dexmedetomidine Different Doses as Adjuvant to Entropy-assisted General Anesthesia During Functional Endoscopy Sinus Surgery. A Randomized Comparative Study
Brief Title: Dexmedetomidine Different Doses as Adjuvant to Entropy-assisted General Anesthesia During Functional Endoscopy Sinus Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Youssef Ollaek, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ms-393-2020
Record Dates: First submitted 2022-01-06; First posted 2022-02-07 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Pain Management; Dexmedetomidine; Anesthesia
Keywords: Entropy; FESS
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G0.2 (Active Comparator): (33) patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minutes followed by infusion at the rate of 0.2 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine
- G0.4 (Active Comparator): (33) patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minutes followed by infusion at the rate of 0.4 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine
- G0.6 (Active Comparator): (33) patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minutes followed by infusion at the rate of 0.6 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minute followed by infusion

SUMMARY:
The aim of work to assess the effect of different doses of Dexmedetomidine when used as an adjuvant to entropy-guided general anesthesia on the intraoperative surgical field quality, inhaled anesthesia consumption and postoperative analgesia requirement during FESS surgeries.

DETAILED DESCRIPTION:
This randomized comparative study is designed to:

* To assess between the effect of different dose Dexmedetomidine infusions on the surgical field quality.
* To determine the effect of different dose of Dexmedetomidine infusions on the required MAC of isoflurane needed to maintain entropy between 40-60.
* To determine the effect of different of Dexmedetomidine on the patient recovery time, and the postoperative analgesic requirement.

Hypothesis

The primary objective of this study is to find out the optimum infusion dose of Dexmedetomidine for the best surgical field quality, reduces inhalational anesthetic requirement without affecting recovery time.

On arrival to the operating room, an 18G cannula will be inserted and 500 ml Ringer acetate solution will be started slowly. Standard monitoring (electrocardiography, pulse oximetry and non-invasive blood pressure monitoring) will be connected to the patient, baseline blood pressure and heart rate will be measured and recorded. The 3-electrode sensor of the entropy (GE carestation 650) will be applied to the patient's forehead and the baseline state entropy (SE) and response entropy (RE) will be recorded. The patient will be premedicated with intravenous Ranitidine 50 mg and Metoclopramide 10 mg. Patients will be equally divided into three equal groups and will be given the following according to group allotted.

G0.2: (33) patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minutes followed by infusion at the rate of 0.2 mcg/kg/hour G0.4: (33) patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minutes followed by infusion at the rate of 0.4 mcg/kg/hour G0.6: (33) patients will receive after induction of anesthesia DEX at 1 mcg/kg for 10 minutes followed by infusion at the rate of 0.6 mcg/kg/hour

Induction of general anesthesia will be carried out using fentanyl 2mcg/kg Propofol 1.5-2 ml/kg and endotracheal intubation will be facilitated with Atracurium 0.5mg/kg.

General anesthesia will be maintained using isoflurane, the vol % will be adjusted at 1.2% to 2% to maintain a target entropy 40-60. The repeated doses of Atracurium 0.1 mg/kg every 20-30 minutes will be administered guided by peripheral nerve stimulator.

Hemodynamics including mean arterial blood pressure and heart rate along with entropy will be recorded every 5 minutes for the first 20 minutes after induction of GA and every 15 minutes till the end of surgery. Bradycardia (Heart rate < 50 beat/min) will be treated with atropine 0.02 mg/kg. Hypotension (MAP < 55 mmHg) will be treated with fluids and Ephedrine 5mg iv. All surgeries will be accomplished by the same surgeon using the same surgical technique. The surgical field quality will be rated by the surgeon once the surgery started and every 30 minutes using a 6-point scale for evaluation of operative field visibility (Boezaart Surgical Field Grading Scale).

Grade Assessment 0 No bleeding (cadaveric conditions)

1. Slight bleeding - no suctioning required
2. Slight bleeding - occasional suctioning required
3. Slight bleeding - frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed
4. Moderate bleeding - frequent suctioning required and bleeding threatens surgical field directly after suction is removed
5. Severe bleeding - constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely compromised

The lowest isoflurane vol % needed to keep a target of 40-60 reading on entropy recorded on the same time table used for the vital signs measured throughout the study. 1 gm of paracetamol will be give intra-venous at the end of surgery.The residual effect of the muscle relaxant will be reversed with administration of neostigmine 0.05 mg/kg and atropine 0.02 mg/kg once TOF count is 2/4. When the patients is able to obey verbal commands, endotracheal tube will be removed after suctioning the airway under direct vision, the patient will then moved to the Post Anesthesia Care Unit (PACU). The recovery time (between stopping of inhalational anesthesia till time of patient obeying) and the duration of Anesthesia defined as time interval between induction of Anesthesia and endotracheal extubation will both calculated and recorded.

Upon arrival to PACU, patients will be monitored with non-invasive blood pressure and pulse oximeter. Oxygen masks will placed on the patients with a flow rate of 6 L/min. The pain will be assessed using the visual analogue scale, and sedation will be assessed using the Ramsay sedation scale every thirty-minutes for two hours. Rescue analgesia will be provided with Pethidine 0.5mg/kg intravenously for those who complained of pain or with VAS score greater than 3.

After two hours, patients that have a score of nine or more on the modified Aldrete discharge scoring system will be discharged to the ward.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) Class I or II undergoing elective functional endoscopic sinus surgery.

Exclusion Criteria:

* American Society of Anaesthesiology (ASA) Class ≥ III
* Allergy or hypersensitivity to Dexamedetomidine.
* History of myocardial dysfunction.
* Cardiac dysrhythmia and Heart block
* Patients receiving beta blockers or calcium channel blockers
* Patient refusal
* Patient with known history of hepatic or renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Surgical field quality using Fromme et al 6-point bleeding scale | Through operative time, an average of 1 to 2 hours
  0 No bleeding (cadaveric conditions)
  1. Slight bleeding - no suctioning required
  2. Slight bleeding - occasional suctioning required
  3. Slight bleeding - frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed
  4. Moderate bleeding - frequent suctioning required and bleeding threatens surgical field directly after suction is removed
  5. Severe bleeding - constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely compromised

SECONDARY OUTCOMES:
Intraoperative hemodynamics including MAP (mmHg) | Through operative time, an average of 1 to 2 hours
  MAP: Mean arterial pressure HR: Heart rate
Intraoperative hemodynamics including HR ( beats/min.) | Through operative time, an average of 1 to 2 hours
  HR: Heart Rate
End tidal isoflurane concentration needed to maintain SE 40-60 | Through operative time, an average of 1 to 2 hours
  SE: State Entropy
  Entropy is a quantitative EEG device which captures a single-lead frontal EEG via a 3-electrode sensor applied to the patient's forehead. The state entropy (SE) scale ranges from 0 (no brain activity) to 91 (fully awake)
End tidal isoflurane concentration needed to maintain RE 40-60 | Through operative time, an average of 1 to 2 hours
  RE: Response Entropy
  Entropy is a quantitative EEG device which captures a single-lead frontal EEG via a 3-electrode sensor applied to the patient's forehead. The response entropy (RE) scale ranges from 0 (no brain activity) to 100 (fully awake).
The duration of anesthesia and recovery time | Through operative and recovery time, an average of 3 to 4 hours
  Duration of Anesthesia: Time interval between induction if Anesthesia and endotracheal extubation.
  The recovery time: Time interval between discontinuation of the inhalational anesthesia and extubation of endotracheal tube.
Postoperative Pain Score | Two hours
  Pain Score: Visual analog scale subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Postoperative Sedation Score | Two hours
  Sedation Score: Ramesy Sedation Scale
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response
Immediate postoperative pethidine consumption (mg) in PACU | Two hours
  PACU: Poat Anesthesia Care Unit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided